CLINICAL TRIAL: NCT02248207
Title: Management of Parkinson's Disease Patients at Their First Visits in a Neurological Practice
Brief Title: Tolerability of Sifrol® in Ambulatory Patients Suffering From Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 248.527
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Parkinson Disease patients
  Interventions: Drug: Pramipexole

INTERVENTIONS:
Drug: Pramipexole
  Other Names: Sifrol®

SUMMARY:
Study to obtain information about the co-operation of the different physician-colleagues in the treatment of patients with Parkinson's disease, both in private practices and clinics and about the primary treatment strategies in the pharmacotherapy of Parkinson's disease and to collect data on the tolerability of Sifrol® in ambulatory patients suffering from Parkinson's disease under routing conditions

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's disease who present to the specialist neurologist practice for the first time without or with referral and who are planned to receive or either be switched to Sifrol or continue the previously prescribed therapy with Sifrol® can be included in this observational study

Exclusion Criteria:

* Neurologists are asked to consider the Summary of Product Characteristics (SPC) for Sifrol®

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Parkinson's disease recruited at specialist neurologist (private practices and clinics)
Sampling Method: Non-Probability Sample
Enrollment: 1293 (Actual)
Dates: Start 2003-01; Primary Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Global Assessment of efficacy by investigator on a 4-point scale | after 8 weeks
Change from Baseline in actual Parkinson symptoms | Baseline, after 8 weeks
Global Assessment of tolerability by investigator on a 4-point scale | after 8 weeks

SECONDARY OUTCOMES:
Number of patients with adverse drug reactions | up to 8 weeks